CLINICAL TRIAL: NCT06486701
Title: Effect of Singing on Vital Signs, Pain, Anxiety in Abdominal Surgery Patients
Brief Title: Effect of Singing in Abdominal Surgery Patients
Acronym: singing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, SEMRA BÜLBÜLOĞLU, Clinical Assoc. Professor, Istanbul Aydın University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 86.2023fbu
Record Dates: First submitted 2024-05-01; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Abdominal Pain; Anxiety
Keywords: Signign; Anxiety; Pain; Vital signs; Abdominal surgery patients
MeSH Terms: conditions — Abdominal Pain; Anxiety Disorders; Pain | interventions — Singing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Singing
  Interventions: Behavioral: have a sing
- No intervention (No Intervention): Control

INTERVENTIONS:
Behavioral: have a sing — Singing
  Other Names: Singing
  Arms: Experimental

SUMMARY:
Patients who have undergone abdominal surgery are given a prompt in the postoperative period and asked to sing the song they remember. Vital signs, pain and anxiety levels are measured before and after singing.

DETAILED DESCRIPTION:
This study is of a randomized controlled type. Patients who have undergone abdominal surgery are divided into experimental and control groups in the early postoperative period. No intervention is made to the control group by the researchers. Vital signs, pain and anxiety levels are measured half an hour apart as pre-test and post-test.

Patients in the experimental group are given a prompt in the postoperative period and asked to sing the song they remember. Pre-test before singing and post-test after singing, vital signs, pain and anxiety levels are measured. It is expected that singing will calm patients, stabilize their vital signs, and reduce anxiety and pain.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal surgery patiens
* 18 and more than age

Exclusion Criteria:

* No abdominal surgery patients
* under 18 age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Vital signs, pain and anxiety: Measurement will be made with the Vital signs, pain and anxiety | total of six month
  It will be measure to sing a song after Abdominal Surgery

SECONDARY OUTCOMES:
Vital signs, pain and anxiety: Measurement will be made with the Vital signs, pain and Anxiety | total of six month
  No intervention, the control group abdominal surgery patients

CONTACTS AND LOCATIONS:
Locations (1):
- Medicana Kadikoy Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No